CLINICAL TRIAL: NCT00538135
Title: BOSCOT: A Randomised Control Trial of Cognitive Behavioural Therapy Plus Treatment as Usual Versus Treatment as Usual in the Treatment of Borderline Personality Disorder
Brief Title: BOSCOT : A Randomised Controlled Trial of Cognitive Behavioural Therapy in Borderline Personality Disorder
Acronym: BOSCOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Wellcome Trust (Other); University of Glasgow (Other); University of London (Other); University of York (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 064027/Z/01/Z
Record Dates: First submitted 2007-09-29; First posted 2007-10-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Borderline Personality Disorder
Keywords: randomised controlled trial; borderline personality disorder; cognitive behavioural therapy; treatment as usual
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive Behaviour Therapy plus Treatment as Usual (CBT plus TAU) for borderline personality disorder.
  CBT is a structured, time limited, psycho-social intervention developed to treat Cluster B personality disorder. Patients are encouraged to engage in treatment through a formulation of their problems within a cognitive framework. Interventions focus on the patient's beliefs and behaviour that impair social and adaptive functioning. Thirty sessions of CBT over one year, each lasting up to one hour, are required to work on long-standing problems and develop new ways of thinking and behaving. Priority is given to behaviours that cause harm to self or others. In addition, participants received the usual treatment they would have received if the trial had not been in place
  Interventions: Behavioral: Cognitive Behavioural Therapy; Other: Treatment as usual
- 2 (Active Comparator): Treatment as Usual.
  All participants received the standard treatment (TAU) they would have received if the trial had not been in place. Although standard treatment may vary across the three sites, and depend on the specific problems of the individual participant, it was thought that all participants would be in contact with mental health services and would have some contact with Accident and Emergency services for repeated self-harm episodes. TAU will be documented carefully after each patient exits the trial.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy
  Arms: 1
Other: Treatment as usual — Standard National Health Service treatment as usual for borderline personality disorder

SUMMARY:
The aim of the study was to investigate if the addition of cognitive behavioural therapy to treatment as usual (CBT plus TAU) in participants with borderline personality disorder would decrease the number of participants with emergency (i.e. unplanned) psychiatric or accident and emergency room contact or episode of deliberate self-harm over twelve months treatment and twelve months follow-up, compared with treatment as usual (TAU). The study also examined whether CBT plus TAU would lead to superior improvement in quality of life, social, cognitive and mental health functioning than TAU alone.

DETAILED DESCRIPTION:
The trial is being carried out in three centres in the UK: Glasgow, London and Ayrshire (Ayrshire and Arran). Treatment as Usual (TAU) therefore reflected what is likely to be available in the UK.

Patients were eligible if they satisfied the following criteria:

1. Aged between 18 and 65.
2. Met criteria for at least 5 items of the borderline personality disorder using the Structured Clinical Interview for DSM IV Axis II Personality Disorders (SCID -II)(First, Gibbon, Spitzer, Williams & Benjamin, 1997)
3. Had received either in-patient psychiatric services or an assessment at Accident and Emergency services or an episode of deliberate self-harm (either suicidal act or self-mutilation) in the previous 12 months.
4. Able to give informed consent.

Exclusion criteria were as follows:

1. Currently receiving in-patient treatment for a mental state disorder,
2. Currently receiving a systematic psychological therapy or specialist service, particularly psychodynamic psychotherapy,
3. Insufficient knowledge of English to enable them to be assessed adequately and to understand the treatment approach,
4. Temporarily resident in the area,
5. The existence of an organic illness, mental impairment, alcohol or drug dependence, schizophrenia or bipolar affective disorder, as assessed by SCID I,/P (W/ Psychotic Screen)(version 2) (First, Spitzer, Gibbon, Williams, 1996).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65.
2. Met criteria for at least 5 items of the borderline personality disorder using the Structured Clinical Interview for DSM IV Axis II Personality Disorders (SCID -II)(First, Gibbon, Spitzer, Williams & Benjamin, 1997)
3. Had received either in-patient psychiatric services or an assessment at Accident and Emergency services or an episode of deliberate self-harm (either suicidal act or self-mutilation) in the previous 12 months.
4. Able to give informed consent.

Exclusion Criteria:

1. Currently receiving in-patient treatment for a mental state disorder,
2. Currently receiving a systematic psychological therapy or specialist service, particularly psychodynamic psychotherapy,
3. Insufficient knowledge of English to enable them to be assessed adequately and to understand the treatment approach,
4. Temporarily resident in the area,
5. The existence of an organic illness, mental impairment, alcohol or drug dependence, schizophrenia or bipolar affective disorder, as assessed by SCID I,/P (W/ Psychotic Screen)(version 2) (First, Spitzer, Gibbon, Williams, 1996).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2002-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the composite outcome of the number of in-patient psychiatric hospitalisations, the number of A& E contacts, and the number of suicidal acts. | At both 12 and 24 months post randomisation.

SECONDARY OUTCOMES:
Secondary outcome measures include the Brief Symptom Inventory, Beck Depression Inventory-II, State-Trait Anxiety Inventory, Social Functioning Questionnaire, Inventory of Interpersonal Problems, Schema Questionnaire (Young), Euro-Qol (EQ-5D) | 6, 12, 18 and 24 months post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Kate Davidson, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Psychological Medicine, Glasgow, Strathclyde, United Kingdom

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793